CLINICAL TRIAL: NCT01250275
Title: Effects of Canola Oil on Blood Vessel Function in Peripheral Arterial Disease (PAD)
Brief Title: Effects of Canola Oil on Blood Vessel Function in Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: St. Boniface Hospital (Other)
Responsible Party: Principal Investigator, Dr. Carla Taylor, Professor, Department of Human Nutritional Sciences, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: B2010:125
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Canola Oil; Peripheral Arterial Disease; Peripheral Vascular Disease; PAD
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases | interventions — Soybean Oil; Coconut Oil; Safflower Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Acute Phase: traditional canola oil (Experimental): Participants will receive banana bread containing traditional canola oil once weekly during the 5-week schedule
  Interventions: Other: traditional canola oil
- Acute Phase: high oleic canola oil (Active Comparator): Participants will receive banana bread containing high oleic canola oil once weekly during the 5-week schedule
  Interventions: Other: high oleic canola oil
- Acute Phase: soybean oil (Active Comparator): Participants will receive banana bread containing soybean oil once weekly during the 5-week schedule
  Interventions: Other: soybean oil
- Acute Phase: high linoleic safflower oil (Active Comparator): Participants will receive banana bread containing high linoleic safflower oil once weekly during the 5-week schedule
  Interventions: Other: high linoleic safflower oil
- Acute Phase: coconut oil (Active Comparator): Participants will receive banana bread containing coconut oil once weekly during the 5-week schedule
  Interventions: Other: coconut oil
- Chronic Phase: traditional canola oil (Experimental): A total of 25 participants with peripheral arterial disease will be assigned foods containing traditional canola oil for a total of 8 weeks
  Interventions: Other: traditional canola oil
- Chronic Phase: safflower oil (Active Comparator): A total of 25 participants with peripheral arterial disease will be assigned foods containing an oil mixture representing the typical western diet for a total of 8 weeks
  Interventions: Other: safflower oil

INTERVENTIONS:
Other: traditional canola oil — Participants (10 healthy and 10 with peripheral arterial disease) will be asked to attend a total of 5 consecutive visits (with a minimum of 6 days between visits) in a fasting state where they will be randomly assigned one food item in the form of banana bread containing 50 gm fat from traditional canola oil.
  Arms: Acute Phase: traditional canola oil
Other: high oleic canola oil — Participants (10 healthy and 10 with peripheral arterial disease) will be asked to attend a total of 5 consecutive visits (with a minimum of 6 days between visits) in a fasting state where they will be randomly assigned one food item in the form of banana bread containing 50 gm fat from high oleic canola oil.
  Arms: Acute Phase: high oleic canola oil
Other: soybean oil — Participants (10 healthy and 10 with peripheral arterial disease) will be asked to attend a total of 5 consecutive visits (with a minimum of 6 days between visits) in a fasting state where they will be randomly assigned one food item in the form of banana bread containing 50 gm fat from soybean oil.
  Arms: Acute Phase: soybean oil
Other: high linoleic safflower oil — Participants (10 healthy and 10 with peripheral arterial disease) will be asked to attend a total of 5 consecutive visits (with a minimum of 6 days between visits) in a fasting state where they will be randomly assigned one food item in the form of banana bread containing 50 gm fat from high linoleic safflower oil.
  Arms: Acute Phase: high linoleic safflower oil
Other: coconut oil — Participants (10 healthy and 10 with peripheral arterial disease) will be asked to attend a total of 5 consecutive visits (with a minimum of 6 days between visits) in a fasting state where they will be randomly assigned one food item in the form of banana bread containing 50 gm fat from coconut oil.
  Arms: Acute Phase: coconut oil
Other: traditional canola oil — Participants with peripheral arterial disease (n=25) will be randomized to daily consumption of food items prepared with traditional canola oil for eight weeks.
  Arms: Chronic Phase: traditional canola oil
Other: safflower oil — Participants with peripheral arterial disease (n=25) will be randomized to daily consumption of foods prepared with an oil mixture representing the typical western diet
  Arms: Chronic Phase: safflower oil

SUMMARY:
The fatty acid composition of canola oil will have beneficial acute and chronic effects on vascular function in individuals with peripheral arterial disease.

DETAILED DESCRIPTION:
Given that much of the evidence for current dietary recommendations for type and amounts of fatty acids is based on heart disease, the proposed research will contribute to the knowledge base for dietary fat recommendations for individuals with established cardiovascular disease. Specifically, this study will establish whether canola oil has positive effects on blood vessel function in individuals with peripheral arterial disease by measuring true clinical endpoints such as ankle-brachial index, walking distance, claudication, and vascular function measures. Additionally, since reduced blood flow contributes to cognitive impairment, this study will explore whether improvements in blood vessel function are also associated with improvements in cognitive function. Given the large proportion of the population affected by atherosclerosis and various forms of cardiovascular disease, there is significant potential for greater consumption and utilization of canola oil if there are beneficial effects on blood vessel function and other indicators of cardiovascular disease risk.

ELIGIBILITY:
Inclusion Criteria:Healthy age-matched participants (acute phase of the study):

* Healthy volunteers, male or female, > 40 years of age;
* Body Mass Index 18-30;
* Glycated hemoglobin <6.5%;
* Fasting serum total cholesterol <4 mmol/L and triglycerides <2.5 mmol/L;
* Blood pressure <140/90 mm Hg;
* Ankle-brachial index of >0.9;
* Willing to comply with the protocol requirements;
* Willing to provide informed consent;
* Participants having completed another food-related study are eligible to participate if it has been more than 3 months since their participation.

Inclusion criteria, peripheral arterial disease participants (acute and chronic phases of the study):

* Male or female, > 40 years of age;
* Documented peripheral arterial disease including those with claudication as defined by an ankle brachial index of ≤0.90 or asymptomatic carotid stenosis of >50%; or who have had a previous intervention for peripheral arterial disease;
* Stable medication profile for the past 3 months with no changes anticipated for the duration of the acute or chronic phases;
* Willing to comply with the protocol requirements;
* Willing to provide informed consent;
* Participants having completed another food study are eligible to participate if it has been more than 3 months since the study was completed.

Exclusion criteria, healthy age-matched participants (acute phase of the study):

* Currently smoking, or smoking within the last 6 months (Note: cigar smoking on an occasional basis will be permitted);
* Presence of a clinically diagnosed disease affecting the heart, liver, kidneys, lungs,gastrointestinal, endocrine or blood/immune systems that requires medical treatment;
* Taking any prescribed medication within the last 3 months with the exception of anti-depressants, birth control and hormone (estrogen) replacement therapy;
* Pregnancy;
* Amputation of upper or lower extremity on both sides;
* Has undergone a surgical procedure requiring local or general anesthetic within the last 3 months;
* History of gastrointestinal reactions or allergies to dietary oils and other ingredients in banana bread such as wheat and eggs;
* Daily consumption of omega-3 supplements.

Exclusion Criteria, Peripheral arterial disease participants (acute and chronic phases of the study):

* Currently smoking, or smoking within the last 6 months (Note: cigar smoking on an occasional basis will be permitted);
* Renal failure requiring dialysis;
* Ongoing cardiovascular event (e.g. angina)or medical illness within the last 3 months;
* Hormone (estrogen) replacement therapy;
* Amputation of leg, foot, arm or hand; post mastectomy or post lymphadenectomy;
* History of gastrointestinal reactions or allergies to dietary oils:for the acute study, to ingredients in banana bread such as wheat and eggs, ang for the chronic study, to one or more ingredients in the study foods which significantly limits the number of study foods that can be consumed;
* Inability to adhere to a regular diet;
* Daily consumption of omega-3 supplements.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Acute study to identify the relative potency of fatty acid compositions on blood vessel function in healthy participants and individuals with peripheral arterial disease. | weekly testing for 5 weeks
  Participants (n=20,10 peripheral arterial disease/10 healthy) will attend 5 weekly visits and receive one food item (banana bread)at each visit. Assessment of endothelial function at 2-hours post consumption. Blood samples will be collected for plasma triglycerides, glucose, insulin, markers of oxidative stress, vascular function, inflammation, and metabolism. Food intake and physical activity will be recorded the day before their first test visit, and the same (foods and activities) will be repeated before each visit. Ankle Brachial Index and Pulse Wave Velocity testing will be done.

SECONDARY OUTCOMES:
To test the effects of canola oil consumption for its effects on vascular function and cardiovascular risk factors in a chronic 8-week study in individuals with peripheral arterial disease. | baseline and at 8 weeks
  Participants (n=50,peripheral arterial disease) will be randomly assigned (25 per group) to food items containing either traditional canola oil or an oil mixutre representing the Western diet. Assessments of vascular function, cognitive function, blood lipid profile, glycated hemoglobin, biomarkers of vascular function, inflammation, oxidative stress, immune function, and metabolism, advanced glycated endproducts, and anthropometrics will be completed at baseline and at 8 weeks.
To explore whether improvements in blood vessel function in the chronic 8-week study are also associated with improvements in cognitive function. | baseline and at 8 weeks
  Participants (n=50, 25/group) with peripheral arterial disease will be randomly assigned to receive daily food item(s) containing traditional canola oil or an oil mixture representing the Western diet. Assessment of cognitive function will occur at baseline and at the end of the 8-week study schedule.
4. To assess compliance and tolerability through subjective feedback provided from participants during the chronic 8-week study. | baseline at at 8 weeks
  Participants (n=50, 25/group) with peripheral arterial disease will be randomly assigned to receive a daily food item(s) containing traditional canola oil or an oil mixture representing the Western diet. Compliance and tolerability with food consumption (including side effects) will be assessed from participants' experiences throughout the 8-week study schedule.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Taylor, PhD, Principal Investigator — University of Manitoba
Locations (1):
- IH Asper Clinical Research Insitute, St. Boniface General Hospital, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Johnson GH, Keast DR, Kris-Etherton PM. Dietary modeling shows that the substitution of canola oil for fats commonly used in the United States would increase compliance with dietary recommendations for fatty acids. J Am Diet Assoc. 2007 Oct;107(10):1726-34. doi: 10.1016/j.jada.2007.07.015. PMID 17904932
- [Background] Toth PP. An urgent matter-identifying your patients' cardiovascular risk and improving their outcomes. Atherosclerosis: the underlying disease. J Fam Pract. 2009 Nov;58(11 Suppl Urgent):S19-25. PMID 19891944
- [Background] Poels MM, van Oijen M, Mattace-Raso FU, Hofman A, Koudstaal PJ, Witteman JC, Breteler MM. Arterial stiffness, cognitive decline, and risk of dementia: the Rotterdam study. Stroke. 2007 Mar;38(3):888-92. doi: 10.1161/01.STR.0000257998.33768.87. Epub 2007 Feb 1. PMID 17272780
- [Background] Waldstein SR, Rice SC, Thayer JF, Najjar SS, Scuteri A, Zonderman AB. Pulse pressure and pulse wave velocity are related to cognitive decline in the Baltimore Longitudinal Study of Aging. Hypertension. 2008 Jan;51(1):99-104. doi: 10.1161/HYPERTENSIONAHA.107.093674. Epub 2007 Nov 19. PMID 18025297
- [Background] Aslam F, Haque A, Foody J, Lee LV. Peripheral arterial disease: current perspectives and new trends in management. South Med J. 2009 Nov;102(11):1141-9. doi: 10.1097/SMJ.0b013e3181bb9ab8. PMID 19864983
- [Background] Mukherjee D, Cho L. Peripheral arterial disease: considerations in risks, diagnosis, and treatment. J Natl Med Assoc. 2009 Oct;101(10):999-1008. doi: 10.1016/s0027-9684(15)31066-x. PMID 19860299
- [Background] Carrero JJ, Lopez-Huertas E, Salmeron LM, Baro L, Ros E. Daily supplementation with (n-3) PUFAs, oleic acid, folic acid, and vitamins B-6 and E increases pain-free walking distance and improves risk factors in men with peripheral vascular disease. J Nutr. 2005 Jun;135(6):1393-9. doi: 10.1093/jn/135.6.1393. PMID 15930443
- [Background] Schiano V, Laurenzano E, Brevetti G, De Maio JI, Lanero S, Scopacasa F, Chiariello M. Omega-3 polyunsaturated fatty acid in peripheral arterial disease: effect on lipid pattern, disease severity, inflammation profile, and endothelial function. Clin Nutr. 2008 Apr;27(2):241-7. doi: 10.1016/j.clnu.2007.11.007. Epub 2008 Jan 31. PMID 18237823
- [Background] Al-Qaisi M, Kharbanda RK, Mittal TK, Donald AE. Measurement of endothelial function and its clinical utility for cardiovascular risk. Vasc Health Risk Manag. 2008;4(3):647-52. doi: 10.2147/vhrm.s2769. PMID 18827914
- [Background] Lane HA, Smith JC, Davies JS. Noninvasive assessment of preclinical atherosclerosis. Vasc Health Risk Manag. 2006;2(1):19-30. doi: 10.2147/vhrm.2006.2.1.19. PMID 17319466
- [Background] Simon A, Chironi G, Levenson J. Comparative performance of subclinical atherosclerosis tests in predicting coronary heart disease in asymptomatic individuals. Eur Heart J. 2007 Dec;28(24):2967-71. doi: 10.1093/eurheartj/ehm487. Epub 2007 Oct 29. PMID 17967818
- [Background] Wang X, Keith JC Jr, Struthers AD, Feuerstein GZ. Assessment of arterial stiffness, a translational medicine biomarker system for evaluation of vascular risk. Cardiovasc Ther. 2008 Fall;26(3):214-23. doi: 10.1111/j.1755-5922.2008.00051.x. PMID 18786091
- [Background] Cohn JN, Duprez DA, Grandits GA. Arterial elasticity as part of a comprehensive assessment of cardiovascular risk and drug treatment. Hypertension. 2005 Jul;46(1):217-20. doi: 10.1161/01.HYP.0000165686.50890.c3. Epub 2005 May 2. PMID 15867132
- [Background] Stamatelopoulos K, Karatzi K, Sidossis LS. Noninvasive methods for assessing early markers of atherosclerosis: the role of body composition and nutrition. Curr Opin Clin Nutr Metab Care. 2009 Sep;12(5):467-73. doi: 10.1097/MCO.0b013e32832f0d99. PMID 19571744
- [Background] Zahradka P, Guzman R, Weighell W, Wright B, Baldwin A, Louis S, et al. Increased consumption of legumes improves arterial stiffness in peripheral vascular disease independent of blood pressure, weight and serum cholesterol. Experimental Biology '09, April 18-22, New Orleans, LA 2009.
- [Background] Ciccarone E, Di Castelnuovo A, Salcuni M, Siani A, Giacco A, Donati MB, De Gaetano G, Capani F, Iacoviello L; Gendiabe Investigators. A high-score Mediterranean dietary pattern is associated with a reduced risk of peripheral arterial disease in Italian patients with Type 2 diabetes. J Thromb Haemost. 2003 Aug;1(8):1744-52. doi: 10.1046/j.1538-7836.2003.00323.x. PMID 12911588
- [Background] Gimeno SG, Hirai AT, Harima HA, Kikuchi MY, Simony RF, de Barros N Jr, Cardoso MA, Ferreira SR; Japanese-Brazilian Diabetes Study Group. Fat and fiber consumption are associated with peripheral arterial disease in a cross-sectional study of a Japanese-Brazilian population. Circ J. 2008 Jan;72(1):44-50. doi: 10.1253/circj.72.44. PMID 18159098
- [Background] Lane JS, Magno CP, Lane KT, Chan T, Hoyt DB, Greenfield S. Nutrition impacts the prevalence of peripheral arterial disease in the United States. J Vasc Surg. 2008 Oct;48(4):897-904. doi: 10.1016/j.jvs.2008.05.014. Epub 2008 Jun 30. PMID 18586439
- [Background] Katsouyanni K, Skalkidis Y, Petridou E, Polychronopoulou-Trichopoulou A, Willett W, Trichopoulos D. Diet and peripheral arterial occlusive disease: the role of poly-, mono-, and saturated fatty acids. Am J Epidemiol. 1991 Jan;133(1):24-31. doi: 10.1093/oxfordjournals.aje.a115798. PMID 1983895
- [Background] Madden J, Brunner A, Dastur ND, Tan RM, Nash GB, Rainger GE, Shearman CP, Calder PC, Grimble RF. Fish oil induced increase in walking distance, but not ankle brachial pressure index, in peripheral arterial disease is dependent on both body mass index and inflammatory genotype. Prostaglandins Leukot Essent Fatty Acids. 2007 Jun;76(6):331-40. doi: 10.1016/j.plefa.2007.04.003. Epub 2007 Jun 27. PMID 17600695
- [Background] Goodfellow J, Bellamy MF, Ramsey MW, Jones CJ, Lewis MJ. Dietary supplementation with marine omega-3 fatty acids improve systemic large artery endothelial function in subjects with hypercholesterolemia. J Am Coll Cardiol. 2000 Feb;35(2):265-70. doi: 10.1016/s0735-1097(99)00548-3. PMID 10676668
- [Background] Hill AM, Buckley JD, Murphy KJ, Howe PR. Combining fish-oil supplements with regular aerobic exercise improves body composition and cardiovascular disease risk factors. Am J Clin Nutr. 2007 May;85(5):1267-74. doi: 10.1093/ajcn/85.5.1267. PMID 17490962
- [Background] Dyerberg J, Eskesen DC, Andersen PW, Astrup A, Buemann B, Christensen JH, Clausen P, Rasmussen BF, Schmidt EB, Tholstrup T, Toft E, Toubro S, Stender S. Effects of trans- and n-3 unsaturated fatty acids on cardiovascular risk markers in healthy males. An 8 weeks dietary intervention study. Eur J Clin Nutr. 2004 Jul;58(7):1062-70. doi: 10.1038/sj.ejcn.1601934. PMID 15220949
- [Background] Nestel P, Shige H, Pomeroy S, Cehun M, Abbey M, Raederstorff D. The n-3 fatty acids eicosapentaenoic acid and docosahexaenoic acid increase systemic arterial compliance in humans. Am J Clin Nutr. 2002 Aug;76(2):326-30. doi: 10.1093/ajcn/76.2.326. PMID 12145002
- [Background] Hjerkinn EM, Abdelnoor M, Breivik L, Bergengen L, Ellingsen I, Seljeflot I, Aase O, Ole Klemsdal T, Hjermann I, Arnesen H. Effect of diet or very long chain omega-3 fatty acids on progression of atherosclerosis, evaluated by carotid plaques, intima-media thickness and by pulse wave propagation in elderly men with hypercholesterolaemia. Eur J Cardiovasc Prev Rehabil. 2006 Jun;13(3):325-33. doi: 10.1097/01.hjr.0000209817.28444.fb. PMID 16926660
- [Background] Rizza S, Tesauro M, Cardillo C, Galli A, Iantorno M, Gigli F, Sbraccia P, Federici M, Quon MJ, Lauro D. Fish oil supplementation improves endothelial function in normoglycemic offspring of patients with type 2 diabetes. Atherosclerosis. 2009 Oct;206(2):569-74. doi: 10.1016/j.atherosclerosis.2009.03.006. Epub 2009 Mar 19. PMID 19394939
- [Background] Murphy KJ, Meyer BJ, Mori TA, Burke V, Mansour J, Patch CS, Tapsell LC, Noakes M, Clifton PA, Barden A, Puddey IB, Beilin LJ, Howe PR. Impact of foods enriched with n-3 long-chain polyunsaturated fatty acids on erythrocyte n-3 levels and cardiovascular risk factors. Br J Nutr. 2007 Apr;97(4):749-57. doi: 10.1017/S000711450747252X. PMID 17349088
- [Background] O'Keefe JH Jr, Abuissa H, Sastre A, Steinhaus DM, Harris WS. Effects of omega-3 fatty acids on resting heart rate, heart rate recovery after exercise, and heart rate variability in men with healed myocardial infarctions and depressed ejection fractions. Am J Cardiol. 2006 Apr 15;97(8):1127-30. doi: 10.1016/j.amjcard.2005.11.025. Epub 2006 Mar 3. PMID 16616012
- [Background] Nicholls SJ, Lundman P, Harmer JA, Cutri B, Griffiths KA, Rye KA, Barter PJ, Celermajer DS. Consumption of saturated fat impairs the anti-inflammatory properties of high-density lipoproteins and endothelial function. J Am Coll Cardiol. 2006 Aug 15;48(4):715-20. doi: 10.1016/j.jacc.2006.04.080. Epub 2006 Jul 24. PMID 16904539
- [Background] Keogh JB, Grieger JA, Noakes M, Clifton PM. Flow-mediated dilatation is impaired by a high-saturated fat diet but not by a high-carbohydrate diet. Arterioscler Thromb Vasc Biol. 2005 Jun;25(6):1274-9. doi: 10.1161/01.ATV.0000163185.28245.a1. Epub 2005 Mar 17. PMID 15774905
- [Background] Fuentes F, Lopez-Miranda J, Sanchez E, Sanchez F, Paez J, Paz-Rojas E, Marin C, Gomez P, Jimenez-Pereperez J, Ordovas JM, Perez-Jimenez F. Mediterranean and low-fat diets improve endothelial function in hypercholesterolemic men. Ann Intern Med. 2001 Jun 19;134(12):1115-9. doi: 10.7326/0003-4819-134-12-200106190-00011. PMID 11412051
- [Background] Nestel PJ, Pomeroy SE, Sasahara T, Yamashita T, Liang YL, Dart AM, Jennings GL, Abbey M, Cameron JD. Arterial compliance in obese subjects is improved with dietary plant n-3 fatty acid from flaxseed oil despite increased LDL oxidizability. Arterioscler Thromb Vasc Biol. 1997 Jun;17(6):1163-70. doi: 10.1161/01.atv.17.6.1163. PMID 9194769
- [Background] Ros E, Nunez I, Perez-Heras A, Serra M, Gilabert R, Casals E, Deulofeu R. A walnut diet improves endothelial function in hypercholesterolemic subjects: a randomized crossover trial. Circulation. 2004 Apr 6;109(13):1609-14. doi: 10.1161/01.CIR.0000124477.91474.FF. Epub 2004 Mar 22. PMID 15037535
- [Background] West SG, Hecker KD, Mustad VA, Nicholson S, Schoemer SL, Wagner P, Hinderliter AL, Ulbrecht J, Ruey P, Kris-Etherton PM. Acute effects of monounsaturated fatty acids with and without omega-3 fatty acids on vascular reactivity in individuals with type 2 diabetes. Diabetologia. 2005 Jan;48(1):113-22. doi: 10.1007/s00125-004-1600-7. Epub 2004 Dec 29. PMID 15624100
- [Background] Cortes B, Nunez I, Cofan M, Gilabert R, Perez-Heras A, Casals E, Deulofeu R, Ros E. Acute effects of high-fat meals enriched with walnuts or olive oil on postprandial endothelial function. J Am Coll Cardiol. 2006 Oct 17;48(8):1666-71. doi: 10.1016/j.jacc.2006.06.057. Epub 2006 Sep 26. PMID 17045905
- [Background] Hall WL. Dietary saturated and unsaturated fats as determinants of blood pressure and vascular function. Nutr Res Rev. 2009 Jun;22(1):18-38. doi: 10.1017/S095442240925846X. Epub 2009 Feb 26. PMID 19243668